CLINICAL TRIAL: NCT06411977
Title: Multiband-/-Bracket Induced Qualitative and Quantitative Changes in the Oral Microbiome and Its Influence by Preventive Intervention Using Dietary Supplements
Brief Title: Effect of Dietary Supplements on the Oral Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Center of Dental Medicine Switzerland (Other)
Collaborators: University of Wuerzburg (Other); Helmholtz Centre for Infection Research (Other)
Responsible Party: Principal Investigator, Dr. Elisabeth Reichardt, Principal Investigator, University Center of Dental Medicine Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01896
Record Dates: First submitted 2024-05-02; First posted 2024-05-14 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Nutrition, Healthy
MeSH Terms: interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Orthodontic patients with fixed appliances
- Juice group (Other): Orthodontic patients with fixed appliances with daily administration of vegetable juice up to 14 days
  Interventions: Dietary Supplement: Vegetable juice

INTERVENTIONS:
Dietary Supplement: Vegetable juice — Vegetable juice (Fa. Fitrabbit, Voglsam)
  Arms: Juice group

SUMMARY:
The oral cavity's microbiome is a diverse community, hosting over 700 bacterial species. Due to its varied niches, the oral cavity constitutes a highly complex environment where different microbes preferentially colonize distinct habitats.

The aim of the study was to investigate the alteration of the oral microbiome during therapy with fixed orthodontic appliances using dietary supplements.

DETAILED DESCRIPTION:
In the randomized clinical trial, the effect of dietary supplements (vegetable juice) was investigated in patients treated with fixed orthodontic appliances. Saliva, tongue and subgingival samples were taken from each participant at three different time points: TO (before insertion of fixed orthodontic therapy), T1 14 days after daily administration of lettuce juice; T2 up to 6 months after washout. Orthodontic patients without dietary intervention served as controls. In addition, clinical indices were examined. Samples were analyzed by Illumina 16S rRNA sequencing and taxonomically assigned.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 12 to 99 years
* Good general condition, healthy
* Inflammation-free marginal periodontium
* Metal brackets in the upper and lower jaw

Exclusion Criteria:

* History of allergies
* Self reported as being immunocompromised
* Self-reported as pregnant or nursing
* Self-reported serious medical conditions
* Antibiotic or anti-inflammatory medication within 6 months before screening visit
* Smoker

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Investigation of gingival indices using Plaque Index (PI) | Baseline (before insertion of fixed orthodontic appliances) T0, two weeks after insertion of orthodontic appliances (T1), 3 months-6 months after baseline (T2)
  To evaluate the plaque-reducing effect of vegetable juice in orthodontic patients in the upper and lower jaw. This index ascertains the thickness of plaque along the gingival margin (Sore 0-3); 0: No plaque 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. 2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Investigation of gingival indices using Periodontal Screening Index (PSI). | Baseline (before insertion of fixed orthodontic appliances) T0, two weeks after insertion of orthodontic appliances (T1), 3 months-6 months after baseline (T2)
  To evaluate the effect of vegetable juice on the periodontal tissues in orthodontic patients in the upper and lower jaw (Score 0-4). 0: Healthy; 1: Bleeding on probing 2: Calculus 3: Dental pocket > 3.5 mm 4: Dental pocket > 5.5 mm
Investigation of gingival indices using Sulcus Bleeding Index. | Baseline (before insertion of fixed orthodontic appliances) T0, two weeks after insertion of orthodontic appliances (T1), 3 months-6 months after baseline (T2)
  To evaluate the inflammation-reducing effect of vegetable juice in orthodontic patients in the upper and lower jaw by counting bleeding on probing from tooth 17 to tooth 47 (Bleeding: yes, No bleeding: no)
To count the number of bacterial colonization on tongue using next-generation-sequencing of the bacterial 16S rRNA gene. | Baseline (before insertion of fixed orthodontic appliances) T0, two weeks after insertion of orthodontic appliances (T1), 3 months-6 months after baseline (T2)
  To determine abundance up to genus level of bacteria in tongue samples in the intervention group (juice group) compared to control group using next-generation-sequencing.
To count the number of bacterial colonization in plaque using next-generation-sequencing of the bacterial 16S rRNA gene. | Baseline (before insertion of fixed orthodontic appliances) T0, two weeks after insertion of orthodontic appliances (T1), 3 months-6 months after baseline (T2)
  To determine abundance up to genus level of bacteria in plaque samples in the intervention group (juice group) compared to control group using next-generation-sequencing.
To count the number of bacterial colonization in saliva using next-generation-sequencing of the bacterial 16S rRNA gene. | Baseline (before insertion of fixed orthodontic appliances) T0, two weeks after insertion of orthodontic appliances (T1), 3 months-6 months after baseline (T2)
  To determine abundance up to genus level of bacteria in saliva in the intervention group (juice group) compared to control group using next-generation-sequencing.

CONTACTS AND LOCATIONS:
Locations (2):
- University of Wuerzburg, Würzburg, Germany
- University Center for Dental Medicine, Basel, Switzerland